CLINICAL TRIAL: NCT03472391
Title: Physical Therapy for In-patients With Severe Anorexia Nervosa: A Randomized Feasibility Study
Brief Title: Physical Therapy for In-patients With Severe Anorexia Nervosa
Acronym: PTSAN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Odense University Hospital (Other)
Collaborators: University of Southern Denmark (Other)
Responsible Party: Principal Investigator, René Klinkby Støving, Professor, Odense University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PTSAN
Record Dates: First submitted 2018-03-06; First posted 2018-03-21 (Actual); Last update posted 2019-03-20 (Actual); Status verified 2019-03

CONDITIONS: Anorexia Nervosa
MeSH Terms: conditions — Anorexia Nervosa | interventions — Physical Therapy Modalities

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Active Comparator): Supervised exercise therapy by physical therapist: patients allocated to physical therapy will participate in a 4-week (2 sessions a week of 40 minutes) supervised and tailored exercise program mainly consisting of light strength training. The exercise program is an add-on treatment to the primary treatment of re-nutrition and somatic stabilization.
  Interventions: Behavioral: Physical Therapy
- Control (No Intervention): The control group follows ordinary treatment in consisting of re-nutrition and somatic stabilization

INTERVENTIONS:
Behavioral: Physical Therapy — A 4-week (2 exercise session af week, of 40 minutes )tailored physiotherapeutic exercise program. The sessions are individually and supervised by physical therapist and tailored to patients with severe anorexia nervosa. The exercise program mainly consist of strength training exercises without any equipment other than a floor mat.
  Arms: Intervention

SUMMARY:
In-patients with severe anorexia nervosa (AN) often drop out of treatment, because of ambivalence towards treatment and anxiety for weight gain. However, physical therapy has shown some positive effects on symptoms of AN. This study aims to investigate the feasibility of a randomized control trial (RCT) of a standardized physiotherapeutic program for patients with severe AN with compliance to nutritional therapy as the primary outcome measure.

DETAILED DESCRIPTION:
Anorexia nervosa (AN) is a serious and complex disease with unknown etiology. It is characterised by disturbed body image and extreme and devastating fear of gaining weight. The illness leads to a considerable and sometimes dangerous weight loss because of the limited food intake and often an exaggerated exercise behavior. AN can affect people of all ages and of both sexes, but girls or young women are more at risk. The prevalence among young women in Denmark is estimated to be between 0.4% and 1%. AN is associated with a high rate of comorbidity and mortality.

The treatment of AN consist of re-feeding and psychotherapy. Different therapeutic methods and theories have been applied, but none have shown to be superior. The patient alliance and motivation for treatment seem to be essential for a successful treatment. Drop-out is a common challenge. Hence, attention must be directed to how the therapeutic alliance and the patient's motivation can be optimized in order to secure a better treatment effect.

Studies have shown that physical therapy, including supervised exercise and bodily focused interventions, may have a positive effect on symptoms of AN. It may reduce the distorted body image and anxiety. However, it is unknown whether physical therapy can affect compliance and drop out rate to the nutrition therapy. The objective of this study is to investigate the feasibility of a RCT design in this group of patients with severe AN at a specialized unit. The intervention is supervised, standardized physical therapeutic exercises mainly consisting of light strength training. The development of the intervention is based partly on the literature, and partly on interviews and observations with two patients with severe AN.

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted to the specialized nutrition section at Odense University Hospital and are fulfilling Diagnostic and Statistical Manual (DSM)-5 criteria for AN.
* 18 years of age or older
* Patients who can be included within the first two weeks of hospitalization

Exclusion Criteria:

* Patients who can not fill in a Danish-language questionnaire.
* Patients who are not able to be in standing position.
* Patients who are not respiratory and circulatory stable.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2017-10-01 (Actual); Primary Completion 2018-05-01 (Actual); Study Completion 2018-05-01 (Actual)

PRIMARY OUTCOMES:
Compliance to overall inpatient treatment. | 4 weeks
  Percentage obtained pre-defined goal weight (0-100%)

SECONDARY OUTCOMES:
Grip strength | Change from baseline to follow-up (4 weeks)
  Grip strength is measured by a hand-held dynamometer. It measures the maximum grip strength force displayed in kilograms.
Functional Movement | Change from baseline to follow-up (4 weeks)
  For assessment of functional movement is the Sit Up Stand Up test (SUSS) used. The test evaluates two functions 1)sit up from supine and 2)squatting form standing position. A score form 0-3 is given (0=poor, 2=intermedium, 3=good).
Quality of Life | Change from baseline to follow-up (4 weeks)
  For assessment of quality of life is the Eating Disorder Quality of Life (EDQoL) questionnaire used.
  EDQLS is a disease-specific quality of life questionnaire developed for use in eating disorders. It consists of 40 items across 12 domains. In each domain patients respond on a 5-point likert scale (strongly agress through strongly disagree). Each domain has three questions, except the eating domain which consists of six questions. The domains are: school/work, family and close relationships, relationships with others, future, feelings, appearance, leisure, values and beliefs, cognitive, physical health, psychological health and eating. Each score is summed using a scoring algorithm with a higher total score indicating higher quality of life (0-200).
Body Image | Change from baseline to follow-up (4 weeks)
  Eating Disorder Inventory (EDI) -3 Danish version is a self-reported assessment with 11 sub-scales, where only one sub-scale is used: body dissatisfaction with 9 items. Answers are given on a 6-point likert scale (highest body dissatisfaction = 6). Total range for the sub-scale: minimum=0 and maximum = 54.
Body Mass Index | Change from baseline to follow-up (4 weeks)
  body weight (kg)/height (m)*height (m)

CONTACTS AND LOCATIONS:
Overall Officials: René K Støving, Principal Investigator — Odense University Hospital
Locations (1):
- Center for eating Disorders, Odense University Hospital, Odense, Denmark

IPD SHARING:
Plan to Share IPD: No